CLINICAL TRIAL: NCT07332143
Title: The Safety and Acceptability of Psilocybin With Support and With Massed Prolonged Exposure Therapy for PTSD
Brief Title: Psilocybin-Assisted Randomized Therapy
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Emory University (Other)
Collaborators: Georgia Department of Veterans Services (Unknown)
Responsible Party: Principal Investigator, Anna Wise, Assistant Professor, Emory University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2025P013649
Record Dates: First submitted 2026-01-08; First posted 2026-01-12 (Actual); Last update posted 2026-01-12 (Actual); Status verified 2026-01

CONDITIONS: PTSD
Keywords: Psilocybin; PTSD; Supportive therapy; PE therapy
MeSH Terms: conditions — Stress Disorders, Post-Traumatic | interventions — Psilocybin; Palliative Care

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Group 1: Psilocybin combined with supportive therapy (Experimental): All participants will receive a single 25 mg dose of psilocybin during the experimental session, which occurs during to their respective therapy model.
  Then, participants will receive 2 support (integrative) therapy sessions that will be 1 week apart. In between these sessions, subjects will complete a series of online surveys to track treatment progress.
  Interventions: Drug: psilocybin; Behavioral: Supportive Therapy
- Group 2: Psilocybin combined with massed prolonged exposure (PE) therapy (Experimental): All participants will receive a single 25 mg dose of psilocybin during the experimental session, followed by 10 prolonged exposure (PE) therapy sessions for 10 days. In between these sessions, participants will complete a series of online surveys to track treatment progress.
  Interventions: Drug: psilocybin; Behavioral: Prolonged Exposure Therapy

INTERVENTIONS:
Drug: psilocybin — 25 mg
  Other Names: 3-[2-(Dimethylamino)ethyl]-1H-indol-4-yl dihydrogen phosphate
Behavioral: Supportive Therapy — Treatment includes non-directive psychological support across the preparatory, dosing, and integration sessions. Preparatory sessions include psychoeducation regarding psilocybin's subjective effects and establish strategies for psilocybin related support, including boundaries around physical touch. Therapists encourage setting intention for dosing day, and practicing experiential exercises. Integration sessions include processing the participant's experience of their psilocybin administration session. Therapists will support participants in identifying activities for ongoing integration outside of sessions. The standard care for supportive therapy will be modeled in this study.
  Arms: Group 1: Psilocybin combined with supportive therapy
Behavioral: Prolonged Exposure Therapy — Prolonged Exposure (PE) Therapy will be conducted for 10 sessions. They will consist of repeated exposures to trauma memories (imaginal exposure) consistent with the manualized protocol for massed exposure therapy. Also consistent with this treatment manual, participants will listen to imaginal exposures and conduct in real life exposures outside of PE sessions for "homework". The standard care for PE therapy will be modeled in this study.
  Arms: Group 2: Psilocybin combined with massed prolonged exposure (PE) therapy

SUMMARY:
This pilot study will examine the safety, tolerability, acceptability, and efficacy of combination psilocybin + psychotherapy to decrease PTSD symptoms. Participants will be randomized into two different treatment groups, allowing the investigators to directly compare PE augmented with psilocybin and psilocybin-assisted psychotherapy.

DETAILED DESCRIPTION:
The Primary objective is to pilot and investigate tolerability, safety, and acceptability of psilocybin-assisted supportive therapy and psilocybin-assisted massed prolonged exposure (PE) therapy and conduct exploratory analyses related to comparative effectiveness of these treatments, including preliminary outcomes from pre-treatment to 1-month follow-up on post-traumatic stress disorder (PTSD) symptoms. Safety and tolerability of the treatment will be assessed and evaluated using the Swiss Psychedelic Side Effects Inventory (SPSI), Psychedelic-assisted Therapy After Effects (PATAE), and the Accessibility Questionnaire (AQ).

The study will also evaluate the effect of psilocybin and massed exposure therapy using Subjective Units of Distress (SUDS) during imaginal exposure sessions; to assess self-reported PTSD and depression symptoms across treatment and investigate effect on fear extinction learning and fear extinction recall as assessed via fear potentiated startle. Given that this is a pilot study with small sample, analyses will be preliminary.

ELIGIBILITY:
Eligible participants must be over the age of 18. They must self-identify as Georgia military veterans, reservists, National Guard members, or active-duty service members. Additionally, they must be seeking treatment for PTSD, which will be confirmed by a CAPS-5-R assessment. The criteria below will be applicable to all participants, regardless of study treatment arm.

Inclusion Criteria

1. Meet criteria for PTSD due to trauma occurring at least 6 months prior based on CAPS-5-R diagnostic scoring rules.
2. Willingness of participant to sign a release for the investigators to communicate with their primary care or mental health providers, if indicated
3. Are 18 years and older.
4. Are able to visually read and understand the English language and give written informed consent.
5. Are able to swallow pills.
6. Agree to have study visits video and/or audio recorded, including dosing session, Independent Rater assessments, and non-drug psychotherapy sessions.
7. Must provide a contact (relative, spouse, close friend, or other support person) who is willing and able to be reached by the investigators in the event of a participant becoming suicidal or unreachable.
8. Must agree to inform the investigators within 48 hours of any medical conditions and procedures.
9. If able to become pregnant, must have a negative pregnancy test prior to study entry, at study entry, and prior to the psilocybin Session. They must agree to use highly effective birth control for a month prior to the psilocybin session and through 10 days after the Medicine session. Highly effective birth control methods include intrauterine device, injected, implanted, intravaginal, or transdermal hormonal methods, abstinence, oral hormones plus a barrier contraception, vasectomized sole partner, or double barrier contraception. Two forms of contraception are required with any barrier method or oral hormones (i.e., condom plus diaphragm, condom or diaphragm plus spermicide, oral hormonal contraceptives plus spermicide or condom). Not able to become pregnant is defined as permanent sterilization, postmenopausal (i.e., 12 consecutive months without menstruation), or assigned male at birth.
10. Agree to the following lifestyle modifications: comply with requirements for fasting and refraining from certain medications prior to the psilocybin Session, not participate in any other interventional clinical trials during the duration of the treatment, and be accompanied to hotel after Medicine Session, and commit to medication dosing, therapy, and study procedures.

Exclusion Criteria

Potential participants are ineligible to enroll in the protocol if they:

1. Are not able to give adequate informed consent.
2. Are currently engaged in compensation litigation whereby financial gain would be achieved from prolonged symptoms of PTSD or any other psychiatric disorders. "Compensation litigation" will not include veterans who are service connected through PTSD or other conditions.
3. Are likely, in the investigator's opinion and via observation during the Preparatory Period, to be re-exposed to their index trauma or other significant trauma, lack social support, or lack a stable living situation.
4. Have any current problem which, in the opinion of the investigator or Medical Monitor, might interfere with participation.
5. Have a family history bipolar disorder type 1 or a psychotic disorder in first degree relatives.
6. Have a history of or current bipolar type 1 disorder, or primary psychotic disorder (e.g., schizophrenia), as assessed via DIAMOND and clinical interview, dementia; or intellectual disability.
7. Have current major depressive disorder with psychotic features assessed via DIAMOND.
8. Have met criteria at any time during their life for hallucinogen substance use disorder.
9. Meet criteria for current (past 3 months) moderate or severe substance use disorder, as defined by 4 or more DSM SUD criteria symptoms.
10. Have a positive screen for cocaine or amphetamines on drug test administered in local community or on site unless being taken as prescribed by a physician.
11. Have current clinically relevant personality pathology.
12. Any participant presenting current serious suicide risk, as determined through psychiatric interview, responses to C-SSRS, and clinical judgment of the investigator will be excluded; however, history of suicide attempts is not an exclusion. Any participant who is likely to require hospitalization related to suicidal ideation and behavior, in the judgment of the investigator, will not be enrolled. Any participant presenting with the following on the C-SSRS administered at screening or baseline will be excluded:

    1. Suicidal ideation score of 4 or greater within the last six months.
    2. Any suicidal behavior, including suicide attempts or preparatory acts, within the last 6 months of the assessment
13. Require ongoing concomitant therapy with a psychiatric medication with exceptions described in protocol section on Concomitant Medications.
14. Other medical exclusion criteria specified in the protocol

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2026-03 (Estimated); Primary Completion 2027-03 (Estimated); Study Completion 2027-03 (Estimated)

PRIMARY OUTCOMES:
Change in PTSD symptoms based on CAPS-5-R total severity score | Baseline, 1-month post-intervention
  PTSD symptoms will be evaluated using the Revised Clinician-Administered PTSD Scale for DSM-5, that refers to 20 core symptoms as CAPS-5, each rated on a 0-4 severity scale (0 = absent to 4 = extremely severe), combining frequency and intensity. Total possible score range is 0 to 80 with higher scores correlating with worse outcome.
Change in PCL-5 score | Baseline, 1, 6 and 12 months post-intervention
  The PCL-5 is a 20-item self-report measure of DSM-5 PTSD symptoms. Scores on the PCL range from 0 to 80, with higher scores indicating higher symptom severity, and a cutoff of 33 indicating clinical levels of PTSD symptoms.
Depression symptoms (PHQ-9) | Baseline, 1, 6 and 12 months post-intervention
  The PHQ-9 is a 9-item self-report measure of depressive symptoms. A score of 10 or above indicative of a possible major depressive episode, and it provides a measure of severity of these symptoms. Total possible score range is 0-29, higher score correlates with worse outcome.

CONTACTS AND LOCATIONS:
Overall Officials: Anna Wise, PhD, Principal Investigator — Emory University
Locations (1):
- Emory University Hospital, Atlanta, Georgia, United States

IPD SHARING:
Plan to Share IPD: No